CLINICAL TRIAL: NCT03978208
Title: A Double-Blind, Placebo-Controlled, Phase 2B Study to Assess the Efficacy and Safety of a 14-Day Dosing Regimen of 3 Doses of ATB-346 Versus Placebo, Orally Administered Once Daily to Patients Diagnosed With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of ATB-346 Versus Placebo in Osteoarthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antibe Therapeutics Inc. (Industry)
Collaborators: Veristat, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATB-346-P2B-DRF
Record Dates: First submitted 2019-03-18; First posted 2019-06-07 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis
Keywords: Knee; WOMAC; NSAID; Pain
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — 2-(6-methoxy-napthalen-2-yl)-propionic acid 4-thiocarbamoyl-phenyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Overencapsulation of study drug tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Comparator (Active Comparator): ATB-346 150 mg overencapsulated tablet taken by mouth once daily for 14 days
  Interventions: Drug: ATB-346 low dose
- ATB-346 mid-dose (Active Comparator): ATB-346 200 mg overencapsulated tablet taken by mouth once daily for 14 days
  Interventions: Drug: ATB-346 mid-dose
- ATB-346 standard dose (Active Comparator): ATB-346 250 mg overencapsulated tablet taken by mouth once daily for 14 days
  Interventions: Drug: ATB-346 standard dose
- Active Comparator (Placebo Comparator): Overencapsulated placebo tablet taken by mouth once daily for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ATB-346 low dose — Double blind comparison of orally administered ATB-346 versus placebo in osteoarthritis patients
  Other Names: Active comparator
  Arms: Placebo Comparator
Other: Placebo — Double blind comparison of orally administered ATB-346 versus placebo in osteoarthritis patients
  Other Names: Non-active comparator
  Arms: Active Comparator
Drug: ATB-346 mid-dose — Double blind comparison of orally administered ATB-346 versus placebo in osteoarthritis patients
  Other Names: Active comparator
  Arms: ATB-346 mid-dose
Drug: ATB-346 standard dose — Double blind comparison of orally administered ATB-346 versus placebo in osteoarthritis patients
  Other Names: Active comparator
  Arms: ATB-346 standard dose

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a 14-day dosing regimen of ATB-346 at doses of 150 mg, 200 mg and 250 mg compared to placebo in reducing osteoarthritis knee pain as measured by changes in the post-treatment WOMAC subscale pain score relative to each patient's pretreatment baseline WOMAC assessment.Safety will be assessed via measurements of vital signs and clinical laboratory tests at baseline and at various time points during the study, patient monitoring, and by the documentation of adverse events.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of a 14-day dosing regimen of once daily administration of ATB-346 at doses of 150 mg, 200 mg and 250 mg compared to placebo in reducing osteoarthritis knee pain as measured by changes in the post-treatment WOMAC subscale pain score relative to each patient's pretreatment baseline WOMAC assessment.A total of 360 evaluable patients are planned in this study: 250 mg (n=120); 200 mg (n=120); 150 mg (n=60); placebo (n=60).

Safety will be assessed via measurements of vital signs and clinical laboratory tests at baseline and at various time points during the study, patient monitoring, and by the documentation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis greater than 2 years duration requiring the use of regular therapies, e.g. oral or topical anti-inflammatories, acetaminophen, topical capsaicin
* Between the ages of 40 to 75
* BMI ≤40
* Patients must be unlikely to procreate or agree to the use of acceptable contraceptive regimens from first drug administration , during the study, and for at least 30 days after the last dose
* Patients must not have used aspirin or naproxen-containing medications for 7 days prior to study entry
* Patients must not have used any anti-inflammatory medications or acetaminophen for 5 days prior to study entry
* Patients must show a ≥10-point increase in WOMAC Visual Analog Score between their screening visit and baseline study entry visit

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Seated and resting pulse rate less than 50 beats per minute (bpm) or more than 100 bpm at screening
* Seated and resting blood pressure below 100/60 mmHg or higher than 140/90 mmHg at screening
* History of significant hypersensitivity to naproxen, other non-steroidal anti-inflammatory agents, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Patients with a history of GI bleeding or ulceration
* Patients refractory to NSAIDs
* Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or know to potentiate or predispose patients to undesired effects
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease as determined by the investigator
* Suicidal tendency, history of/or disposition to seizures, state of confusion
* History of hepatic disease
* Maintenance therapy with any drug, including gastroprotective agents such as proton pump inhibitors, H2 receptor antagonists, sucralfate, etc., or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 30 days before Day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of CYP enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort) in the previous 30 days before Day 1 of this study
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive H. Pylori Urea Breathe Test
* Positive urine screening of alcohol and/or drugs of abuse at the screening visit
* Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAg) or anti-Hepatitis C Virus (HCV) tests
* Females who are pregnant according to a positive serum pregnancy test
* Patients who took an Investigational Product (in another clinical trial) in the previous 30 days before Day 1 of this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
5-item pain intensity measure | Previous 48 hours
  Self reported pain intensity over the past 48 hours. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total between 0 and 50

SECONDARY OUTCOMES:
2-item stiffness intensity measure | Previous 48 hours
  Self reported pain intensity over the past 48 hours. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total between 0 and 20
17-item difficulty performing daily activities measure | Previous 48 hours
  Self reported pain intensity over the past 48 hours. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total between 0 and 170
Measurement of whole blood cyclo-oxygenase activity | After 1, 4 and 14 days of treatment dosing.
  Thromboxane B2 (TXB2) blood levels (pg/mL) will be measured after 1, 4 and 14 days of treatment. samples taken on days 1, 4 and 14. Decreases (measured in pg/mL) in the blood levels of thromboxane B2 are a direct measure of the effect of treatment on cyclo-oxygenase activity and the reduced production of this inflammatory mediator, i.e., thromboxane B2.
Number of patients with genetic variations in the drug modifying enzyme CYP2C9 that may alter the metabolism of ATB-346 will be investigated. | Samples will be retained through study completion and analyzed within 1 year of study initiation.
  CYP2C9 isoforms will be measured in one blood sample taken prior to study drug dosing.
Number of participants with treatment-related adverse events | Pre-study and days 4, 14 and 24.
  The safety of ATB-346 will be monitored via on study and two week post study physician and clinical laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Study Director — Veristat
Locations (35):
- Canada (35):
  - Viable Clinical Research Corp, Mission, British Columbia
  - Ocean West Research Clinic, Surrey, British Columbia
  - James K. Lai MD Inc, Vancouver, British Columbia
  - Dr. MB Jones Inc, Victoria, British Columbia
  - True North Clinical Research Inc., Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Manna Research (Burlington North), Burlington, Ontario
  - Etobicoke Medical Centre, Etobicoke, Ontario
  - Dawson Clinical Research, Guelph, Ontario
  - Dr. Allen Greenspoon Medicine Professional Corporation, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - KGK Science Inc, London, Ontario
  - Malton Medical Clinic, Mississauga, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - King Street Medical Clinic, Oshawa, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Viable Clinical Research Corp, Scarborough Village, Ontario
  - Dr. Steven V. Zizzo Medicine Professional Corporation, Stoney Creek, Ontario
  - Manna Research (Stoney Creek), Stoney Creek, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - LMC Clinical Research Inc, Toronto, Ontario
  - Manna Research (Toronto), Toronto, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Clinical Research& Arthritis Centre, Windsor, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Manna Research (Mirabel QC), Mirabel, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Manna Research (Montreal), Pointe-Claire, Quebec
  - Diex Recherche Quebec Inc., Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Victoriaville Inc., Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: No